CLINICAL TRIAL: NCT01794000
Title: A Phase 3, Double-Blind, Randomized, Efficacy and Safety Comparison of Prasugrel and Placebo in Pediatric Patients With Sickle Cell Disease.
Brief Title: A Study of Prasugrel in Pediatric Participants With Sickle Cell Disease (SCD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study is being terminated for lack of efficacy.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13038; H7T-MC-TADO (Other: Eli Lilly and Company); 2012-003837-41 (EudraCT Number)
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel (Experimental): Participants will be titrated from initial daily dose of 0.08 milligram per kilogram (mg/kg) of orally administered prasugrel monotherapy at randomization to a dose that will achieve a P2Y12 reaction units (PRU) level of 231 to 136, as measured by VerifyNow instrument. This corresponds to a range of platelet inhibition of approximately 30% to 60%. The maximum possible dose allowed is 0.12 mg/kg daily, not to exceed 10 mg daily.
  Interventions: Drug: Prasugrel
- Placebo (Placebo Comparator): Participants in this treatment group will receive daily orally administered placebo and will follow visit schedule identical to that in the active treatment group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prasugrel — Administered orally
  Other Names: LY640315; Effient; Efient
  Arms: Prasugrel
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of the study is to evaluate the efficacy and safety of the study drug known as prasugrel for the reduction of Vaso-Occlusive Crisis events in pediatric participants with sickle cell disease. The study will also investigate reduction in daily pain in children who have sickle cell disease.

DETAILED DESCRIPTION:
The submission database was validated for data reported through the data cutoff date for the submission database lock (SDBL). The SDBL data cutoff was 17 July 2015 for all participants except for 2 in the youngest age group, for whom the SDBL data cutoff occurred on 08 August 2015. The data cutoff date for SDBL corresponds to the primary completion date for the study. The SDBL occurred on 31 August 2015.

The study was stopped following SDBL and review of the topline information indicated that the primary and secondary efficacy endpoints were not met. Subsequently, the Sponsor requested that participants discontinue study drug immediately and that discontinuation visits for all active study participants be conducted as soon as feasible.

After the data cutoff date for SDBL, the Sponsor continued to collect safety data through the final participants contact; some additional efficacy data were collected through the final visit. The last patient visit (LPV) occurred on 17 December 2015, which corresponds to the study completion date and led to the planned supplemental database lock (PSDBL) on 22 January 2016. This supplemental data base was originally designed to capture additional blinded and randomized information to enhance safety data for labeling should the study have been positive.

The safety information contained in this record reflects the entire safety information and reflects the information from the supplemental data base lock in January of 2016. The efficacy information contained in this record reflects the information collected through primary completion date in the submission database. Primary analyses of the major efficacy objectives were repeated using the entire double-blind period data from the PSDBL and did not change the original conclusions and were consistent with the results from the original efficacy analyses included in the SDBL.

ELIGIBILITY:
Inclusion Criteria:

* Have SCD [homozygous sickle cell (HbSS) or hemoglobin (HbS) Beta^0 thalassemia]
* Are participants with SCD who have had ≥2 episodes of vaso-occlusive crisis (VOC) in the past year
* Have a body weight ≥19 kilograms (kg) and are ≥2 and <18 years of age, inclusive at the time of screening
* If participants are ≥2 and ≤16 years of age, must have had a transcranial Doppler within the last year

Exclusion Criteria:

* History of: transient ischemic attack (TIA)/ ischemic or hemorrhagic stroke, severe head trauma, intracranial hemorrhage, intracranial neoplasm, arteriovenous malformation, or aneurysm
* History of abnormal or conditional [velocity in middle or anterior cerebral, or internal carotid artery ≥170 centimeter per second (cm/sec)] transcranial Doppler within the last year
* History of, or are undergoing treatment with, chronic red blood cell (RBC) transfusion therapy
* Are at an increased risk for bleeding complications
* Are receiving chronic treatment with nonsteroidal anti-inflammatory drug (NSAID)s and cannot be switched to another analgesic

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 341 (Actual)
Dates: Start 2013-04; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (50):
- United States (20):
  - Children's Hospital of Oakland, Oakland, California
  - Stanford Univ Medical Center, Palo Alto, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Howard University Hospital, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Childrens Hospital of Michigan, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Albert Einstein College of Medicine, The Bronx, New York
  - University of NC at Chapel Hill School of Medicine, Chapel Hill, North Carolina
  - Childrens Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St Christophers Hospital For Children, Philadelphia, Pennsylvania
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St Jude Childrens Research Hospital, Memphis, Tennessee
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montegnée
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro, Brazil
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec, Canada
- Egypt (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Al Fayyum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Al Mansurah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alexandria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cairo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ismailia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagazig
- Ghana (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Agogo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Korle Bu
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Modena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Verona
- Kenya (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Busia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kisumu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kombewa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nairobi
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beirut, Lebanon
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Muscat, Oman
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeddah, Saudi Arabia
- Turkey (Türkiye) (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Balcali Adana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mersin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Abu Dhabi, United Arab Emirates
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tooting, London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Heeney MM, Hoppe CC, Abboud MR, Inusa B, Kanter J, Ogutu B, Brown PB, Heath LE, Jakubowski JA, Zhou C, Zamoryakhin D, Agbenyega T, Colombatti R, Hassab HM, Nduba VN, Oyieko JN, Robitaille N, Segbefia CI, Rees DC; DOVE Investigators. A Multinational Trial of Prasugrel for Sickle Cell Vaso-Occlusive Events. N Engl J Med. 2016 Feb 18;374(7):625-35. doi: 10.1056/NEJMoa1512021. Epub 2015 Dec 8. PMID 26644172
- See also: A Multinational Trial of Prasugrel for Sickle Cell Vaso-Occlusive Events — http://www.nejm.org/doi/full/10.1056/NEJMoa1512021#t=articleTop

RESULTS

PARTICIPANT FLOW:
Groups:
- Prasugrel: Participants (Pts.) will be titrated from initial daily dose of 0.08 milligram per kilogram (mg/kg) of orally administered prasugrel monotherapy at randomization to a dose that will achieve a P2Y12 reaction units (PRU) level of 231 to 136, as measured by VerifyNow instrument. This corresponds to a range of platelet inhibition of approximately 30% to 60%. The maximum possible dose allowed is 0.12 mg/kg daily, not to exceed 10 mg daily.
Period: Double-Blind Phase (DBP)
Arm/Group | Prasugrel | Placebo
Started | 171 | 170
Received at Least One Dose of Drug | 170 | 170
Discontinued During Double Blind Phase | 169 | 166
Completed | 2 | 4
Not Completed | 169 | 166
Not completed — Adverse Event | 5 | 2
Not completed — Death | 1 | 2
Not completed — Entry Criteria Not Met | 2 | 0
Not completed — Parent/Caregiver Decision | 5 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Sponsor Decision | 148 | 149
Not completed — Withdrawal by Subject | 6 | 11
Period: Open-Label Extension Phase (OLE)
Arm/Group | Prasugrel | Placebo
Started | 3 (Pts. who had not permanently discontinued study drug and concluded DBP were eligible to enter OLE) | 0 (Placebo arm was not applicable to Open-Label Extension Phase)
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Sponsor Decision | 3 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prasugrel | Placebo | Total
Number analyzed (Participants) | 171 | 170 | 341
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.606 (4.334) | 10.580 (4.349) | 10.593 (4.335)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 86 | 173
  Male | 84 | 84 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 94 | 98 | 192
  Unknown or Not Reported | 75 | 71 | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 113 | 109 | 222
  White | 58 | 58 | 116
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 48
  Egypt | 23 | 22 | 45
  United Kingdom | 5 | 4 | 9
  Ghana | 29 | 28 | 57
  Kenya | 47 | 44 | 91
  Oman | 2 | 4 | 6
  Lebanon | 8 | 8 | 16
  Saudi Arabia | 1 | 0 | 1
  Canada | 4 | 4 | 8
  Turkey | 20 | 22 | 42
  Belgium | 1 | 2 | 3
  Brazil | 1 | 0 | 1
  Italy | 7 | 7 | 14
Hydroxyurea Use at Baseline [Number; unit: participants]
  Yes | 77 | 76 | 153
  No | 94 | 94 | 188

OUTCOME MEASURES:

1. Primary Outcome: Number of Vaso-Occlusive Crisis (VOC) Events Per Participant Per Year (Rate of VOC)
Description: The VOC is a composite endpoint of painful crisis or acute chest syndrome. Events that occurred within 7 days from the prior event onset date were not counted as a new episode. Data collected through the primary completion date reported below.
Time Frame: Randomization through 24 Months
Population: All randomized participants.
Measure: Number; unit: Number of Events per Participant-Year
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 171 | 170
Number of Events per Participant-Year | 2.295 | 2.767
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; The time to a recurrent episode of VOC was analyzed using Andersen-Gill model. A robust variance estimate was used, with treatment, hydroxyurea use at baseline and age group included as factors in the model; Test type: Superiority or Other; p = .117, Andersen-Gill model; Rate Ratio = 0.83, 95% CI 2-sided [0.66 to 1.05] — The rate ratio and 2-sided 95% Confidence Interval (CI) were estimated from the Andersen-Gill model

2. Secondary Outcome: Monthly Rate of Days With Pain
Description: Monthly rate of days with pain was measured through participant diaries using a modified version of the Faces Pain Scale-Revised (FPS-R). Each day participants selected the face on the scale that reflected their worst pain related to sickle cell disease (SCD) on that day. This pain scale contains six faces corresponding to the pain intensity of 0, 2, 4, 6, 8 or 10, in which 0 denotes no pain and 10 denotes the worst pain possible. Any day the participant selected a face other than face 0 was considered a day with pain. Monthly rate of days with pain was calculated for each participant by summing the number of days reported with any pain divided by the number of non-missing diary entries completed in the month. A month was defined as 4 weeks (28 days).The monthly rate was set to missing if there were more than 14 missing entries for the FPS-R in a specific month. Data collected through the primary completion date are present below.
Time Frame: Randomization through 9 Months
Population: All randomized participants who are 7 years or older and have both baseline and at least one post-baseline monthly outcome measure in any month. This is the Sickle cell population in which content validity has been established for the FPS-R.
Measure: Least Squares Mean (Standard Error); unit: Percentage of Days in a Month
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 127 | 127
Percentage of Days in a Month | 17.457 (1.558) | 17.699 (1.551)
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; Test type: Superiority or Other; p = .912, Mixed Models Analysis — Mixed Model Repeated Measures (MMRM) included fixed effects of treatment, baseline value of the pain-diary outcome measure, hydroxyurea use, age group, time and treatment-by-time interaction; Least Square Mean Difference = -0.242, 95% CI 2-sided [-4.564 to 4.079] — The Least Square (LS) Mean difference of prasugrel minus placebo and the corresponding 2-sided 95% CI were estimated from the MMRM model

3. Secondary Outcome: Monthly Mean in Faces Pain Scale-Revised Score
Description: Each day participants selected the face on the FPS-R scale that reflected their worst pain related to sickle cell disease (SCD) on that day. Monthly mean in FPS-R score was calculated for each participant by summing the FPS-R score divided by the number of non-missing diary entries completed in the month. This pain scale contains six faces corresponding to the pain intensity of 0, 2, 4, 6, 8 or 10, in which 0 denotes no pain and 10 denotes the worst pain possible. A month was defined as 4 weeks (28 days). The monthly mean in FPS-R score was set to missing if there were more than 14 missing entries for the FPS-R in a specific month. Data collected through the primary completion date are presented below.
Time Frame: Randomization through 9 Months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 127 | 127
Units on a Scale | 0.7116 (0.0757) | 0.6148 (0.0753)
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; Test type: Superiority or Other; p = .365, Mixed Models Analysis — MMRM model included fixed effects of treatment, baseline value of the pain-diary outcome measure, hydroxyurea use, age group, time and treatment-by-time interaction; Least Square Mean Difference = 0.0968, 95% CI 2-sided [-0.1132 to 0.3068] — The LS Mean difference of prasugrel minus placebo and the corresponding 2-sided 95% CI were estimated from the MMRM model

4. Secondary Outcome: Number of Painful Crisis Events Per Participant Per Year (Rate of Painful Crisis)
Description: A painful crisis is defined as an onset of moderate to severe pain that lasts at least 2 hours for which there is no explanation other than vaso-occlusion and which requires therapy with oral or parenteral opioids, ketorolac, or other analgesics prescribed by a health care provider (HCP) in a medical setting such as a hospital, clinic, emergency room visit, or telephone management. The painful crisis that occurred within 7 days from the prior event onset date was not counted as a new episode. Data collected through the primary completion date are presented below.
Time Frame: Randomization through 24 Months
Population: All randomized participants.
Measure: Number; unit: Number of Events per Participant-Year
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 171 | 170
Number of Events per Participant-Year | 2.239 | 2.720
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; Test type: Superiority or Other; p = .109, Andersen-Gill Model — The time to a recurrent episode of painful crisis was analyzed using Andersen-Gill model; A robust variance estimate was used, with treatment, hydroxyurea use at baseline and age group included as factors in the model; Rate Ratio = 0.82, 95% CI 2-sided [0.65 to 1.04] — The rate ratio and 2-sided 95% CI were estimated from the Andersen-Gill model

5. Secondary Outcome: Number of Hospitalizations for VOC Per Participant Per Year (Rate of Hospitalizations)
Description: Hospitalization that occurred within 7 days of the prior event onset date were not counted as a new episode. Data collected through the primary completion date are presented below.
Time Frame: Randomization through 24 Months
Population: All randomized participants.
Measure: Number; unit: Number of Events per Participant-Year
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 171 | 170
Number of Events per Participant-Year | 1.064 | 1.126
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; Test type: Superiority or Other; p = .759, Andersen-Gill model — The time to a recurrent episode of hospitalization was analyzed using Andersen-Gill model; [statistical method as in outcome 4, analysis 1]; Rate Ratio = 0.94, 95% CI 2-sided [0.65 to 1.37] — The rate ratio and 2-sided 95% CI were estimated from the Andersen-Gill model

6. Secondary Outcome: Number of Acute Chest Syndrome Per Participant Per Year (Rate of Acute Chest Syndrome)
Description: Acute chest syndrome was defined as an acute illness characterized by fever and/or respiratory symptoms, accompanied by a new pulmonary infiltrate on a chest X-ray. Acute chest syndrome that occurred within 7 days of the prior event onset date was not counted as a new episode. Data collected through the primary completion date are presented below.
Time Frame: Randomization through 24 Months
Population: All randomized participants.
Measure: Number; unit: Number of Events per Participant-Year
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 171 | 170
Number of Events per Participant-Year | 0.112 | 0.115
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; Test type: Superiority or Other; p = .916, Andersen-Gill model — The time to a recurrent episode of acute chest syndrome was analyzed using Andersen-Gill model; [statistical method as in outcome 4, analysis 1]; Rate Ratio = 0.96, 95% CI 2-sided [0.48 to 1.93] — The rate ratio and 2-sided 95% CI were estimated from the Andersen-Gill model

7. Secondary Outcome: Number of Red Blood Cell (RBC) Transfusions Due to Sickle Cell Disease (SCD) Per Participant Per Year (Rate of RBC Transfusions)
Description: RBC transfusions that occurred within 7 days of the prior event onset date were not counted as a new episode. Data collected through the primary completion date are presented below.
Time Frame: Randomization through 24 Months
Population: All randomized participants.
Measure: Number; unit: Number of Events per Participant-Year
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 171 | 170
Number of Events per Participant-Year | 0.497 | 0.420
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; Test type: Superiority or Other; p = .544, Andersen-Gill model — The time to a recurrent episode of RBC transfusion was analyzed using Andersen-Gill model; [statistical method as in outcome 4, analysis 1]; Rate Ratio = 1.17, 95% CI 2-sided [0.71 to 1.91] — The rate ratio and 2-sided 95% CI were estimated from the Andersen-Gill model

8. Secondary Outcome: Monthly Rate of Days of Analgesic Use
Description: Monthly rate of days of analgesic use was measured through participant diaries and was calculated for each participant by summing the number of days they reported analgesic use divided by the number of diary entries completed in the month. A month was defined as 4 weeks (28 days). The monthly rate was set to missing if there were more than 14 missing entries for analgesic use in a specific month. Data collected through the primary completion date are presented below.
Time Frame: Randomization through 9 Months
Population: All randomized participants who are 4 years or older and have baseline and at least one post-baseline monthly outcome measure in any month. Diaries were only provided to participants 4 years and older.
Measure: Least Squares Mean (Standard Error); unit: Percentage of Days in a Month
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 153 | 153
Percentage of Days in a Month | 24.270 (2.290) | 22.757 (2.337)
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; Test type: Superiority or Other; p = .602, Mixed Models Analysis — The MMRM model included the fixed effects of treatment, the baseline value of the pain-diary measure, hydroxyurea use, age group, time and treatment-by-time interaction; Least Square Mean Difference = 1.513, 95% CI 2-sided [-4.186 to 7.213] — The Least Square Mean difference of prasugrel minus placebo and the corresponding 2-sided 95% CI were estimated from the MMRM model

9. Secondary Outcome: Quarterly Rate of School Absence Due to Sickle Cell Pain
Description: Quarterly rate of school absence due to sickle cell pain was measured through participant diaries and was calculated for each participant by summing the number of days with school absence due to sickle cell pain divided by the number of school dates in the quarter. A quarter was defined as 12 weeks. The quarterly rate was set to missing if there were more than 6 weeks of missing diary entries during a specific quarter. Data collected through the primary completion date are presented below.
Time Frame: Randomization through 9 Months
Population: All Randomized participants who are 4 years or older and have both baseline and at least one post-baseline quarterly outcome measure in any quarter. Diaries were only provided to participants 4 years and older.
Measure: Least Squares Mean (Standard Error); unit: Percentage of Days in a Quarter
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 105 | 115
Percentage of Days in a Quarter | 11.527 (1.525) | 10.255 (1.466)
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; Test type: Superiority or Other; p = .459, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]; Least Square Mean Difference = 1.272, 95% CI 2-sided [-2.109 to 4.652] — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: Time to First Transient Ischemic Attack (TIA)/Ischemic Stroke
Time Frame: Randomization through 24 Months
Population: No participants had a TIA or ischemic stroke at time of analysis.
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Days Hospitalized for VOC
Description: The total length of hospitalization in days for VOC was calculated for each participant. Data collected through the primary completion date are presented below.
Time Frame: Randomization through 24 Months
Population: All randomized participants who were hospitalized for VOC.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 69 | 76
Days | 12.9 (1.72) | 12.0 (1.63)
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; Test type: Superiority or Other; p = .662, ANCOVA — The ANCOVA model included the factors of treatment, hydroxyurea use, age group, and length of follow-up; Least Square Mean Difference = 0.94, 95% CI 2-sided [-3.31 to 5.19] — The LS Mean difference of prasugrel minus placebo and 2-sided 95% CI were estimated from the ANCOVA model

12. Secondary Outcome: Time From Randomization to First and Second VOC
Description: Data collected through the primary completion date are presented below.
Time Frame: Randomization to First VOC and Second VOC respectively (up to 24 Months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 171 | 170
Days
  Time from Randomization to the First VOC | 90.0 [71.0 to 151.0] | 87.0 [65.0 to 106.0]
  Time from Randomization to the Second VOC | 338.0 [240.0 to NA] — Upper limit of 95% Confidence Interval could not be calculated due to limited data | 238.0 [177.0 to 300.0]
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; Time from Randomization to the First VOC; Test type: Superiority or Other; p = .317, Log Rank; A stratified log-rank test were performed with hydroxyurea use and age group as the stratification factors
Statistical Analysis 2: Comparison: Prasugrel vs Placebo; Time from Randomization to the Second VOC; Test type: Superiority or Other; p = .133, Log Rank; A stratified log-rank test were performed with hydroxyurea use and age group as the stratification factors

13. Secondary Outcome: Percentage of Participants With Hemorrhagic Events Requiring Medical Intervention
Description: Medical intervention was defined as any medical evaluation resulting in therapy or further investigation, as determined by a trained medical professional. Data collected from the first dose of study medication through 10 days after last dose of study medication during the double blind study period are presented below.
Time Frame: First Dose through 24 Months
Population: All randomized participants who received at least one dose of drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Prasugrel | Placebo
Number analyzed (Participants) | 170 | 170
Percentage of Participants | 6.5 | 4.7
Statistical Analysis 1: Comparison: Prasugrel vs Placebo; Test type: Superiority or Other; p = .638, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events reported below reflect the entire study safety information through the supplemental data base lock (the study completion date).
Description: All randomized participants who received at least one dose of drug.
Groups:
- Prasugrel - Double Blind Phase: Participants will be titrated from initial daily dose of 0.08 milligram per kilogram (mg/kg) of orally administered prasugrel monotherapy at randomization to a dose that will achieve a P2Y12 reaction units (PRU) level of 231 to 136, as measured by VerifyNow instrument. This corresponds to a range of platelet inhibition of approximately 30% to 60%. The maximum possible dose allowed is 0.12 mg/kg daily, not to exceed 10 mg daily.
- Placebo - Double Blind Phase: Participants in this treatment group will receive daily orally administered placebo and will follow visit schedule identical to that in the active treatment group.
- Prasugrel - Open Label Phase: Participants who continued to meet eligibility criteria, who were not permanently discontinued from study drug, and who concluded their participation in 24 months of double blind treatment were to be considered eligible to enter the open label phase.
Arm/Group | Prasugrel - Double Blind Phase | Placebo - Double Blind Phase | Prasugrel - Open Label Phase
Serious Adverse Events (participants affected / at risk) | 100/170 | 106/170 | 0/3
Other Adverse Events (participants affected / at risk) | 148/170 | 154/170 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Prasugrel - Double Blind Phase (N=170) | Placebo - Double Blind Phase (N=170) | Prasugrel - Open Label Phase (N=3)
Anaemia (Blood and lymphatic system disorders) | 17 (34) | 20 (23) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 0 (0)
Hypersplenism (Blood and lymphatic system disorders) | 3 (4) | 1 (1) | 0 (0)
Intravascular haemolysis (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 75 (187) | 83 (202) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Disorder of orbit (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 5 (6) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic sequestration (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acinetobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis a (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis c (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 11 (12) | 11 (14) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parvovirus b19 infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Plasmodium falciparum infection (Infections and infestations) | 6 (7) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 7 (7) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyomyositis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 4 (4) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Viral tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Serum ferritin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal papillary necrosis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1/87 (1) | 0 (0) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 2/84 (3) | 0 (0)
Thrombosis corpora cavernosa (Reproductive system and breast disorders) | 0 (0) | 1/84 (1) | 0 (0)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 14 (16) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Selective abortion (Surgical and medical procedures) | 1/87 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel - Double Blind Phase (N=170) | Placebo - Double Blind Phase (N=170) | Prasugrel - Open Label Phase (N=3)
Anaemia (Blood and lymphatic system disorders) | 6 (8) | 11 (13) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 90 (223) | 102 (272) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 17 (23) | 20 (28) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 11 (14) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (10) | 12 (16) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 11 (12) | 0 (0)
Gastritis (Gastrointestinal disorders) | 10 (13) | 10 (19) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (11) | 12 (19) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 18 (31) | 19 (30) | 0 (0)
Pyrexia (General disorders) | 35 (54) | 43 (69) | 1 (1)
Malaria (Infections and infestations) | 33 (62) | 33 (53) | 0 (0)
Nasopharyngitis (Infections and infestations) | 15 (19) | 18 (34) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (4) | 10 (11) | 0 (0)
Rhinitis (Infections and infestations) | 11 (12) | 7 (10) | 0 (0)
Tonsillitis (Infections and infestations) | 20 (26) | 24 (31) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 44 (76) | 37 (69) | 0 (0)
Urinary tract infection (Infections and infestations) | 17 (26) | 17 (17) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (11) | 10 (11) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (32) | 29 (54) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 (45) | 47 (84) | 0 (0)
Headache (Nervous system disorders) | 25 (32) | 29 (43) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (19) | 17 (19) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 (48) | 21 (29) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 8 (8) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was stopped following Submission Database Lock, the topline information indicated that the primary and secondary efficacy endpoints were not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days